CLINICAL TRIAL: NCT04092153
Title: A Prospective Randomised Control Trial Comparing Mako Robotic-arm Assisted Functionally Aligned Total Knee Arthroplasty Versus Mako Robotic-arm Assisted Mechanically Aligned Total Knee Arthroplasty
Brief Title: Mako Functionally Aligned Total Knee Arthroplasty vs Mako Mechanically Aligned Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Stryker Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 17/0721
Record Dates: First submitted 2019-09-13; First posted 2019-09-17 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Osteo Arthritis Knee; Osteoarthritis; Surgery
Keywords: total knee arthroplasty; total knee replacement; functional alignment; kinematic alignment; robotic surgery; mako robot; makoplasty; patient outcomes
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Mechanically aligned (Active Comparator): Neutral limb alignment irrespective of the patient's native knee anatomy and joint mechanics
  Interventions: Device: Total knee arthroplasy
- Functionally aligned (Experimental): Restore the patient's own pre-arthritic knee anatomy
  Interventions: Device: Total knee arthroplasy

INTERVENTIONS:
Device: Total knee arthroplasy — Surgical implantation of prosthetic knee using robotic-arm assist

SUMMARY:
This study evaluates outcomes of robotic-arm assisted mechanically aligned total knee arthroplasty [MA TKA] versus robotic-arm assisted functionally aligned total knee arthroplasty [FA TKA]. Half the study will receive MA TKA and half will receive FA TKA.

DETAILED DESCRIPTION:
Total knee arthroplasty [TKA] is an estabilshed treatment for symptomatic end-stage knee osteoarthritis, but there is a higher disatisfaction rate when compared to total hip arthroplasty. The exact aetiology of this is not clear but recent studies have shown one possible reason to be conventional TKA with mechanical alignment [MA] may force the knee into an unnatural position. This may lead to altered knee anatomy and kinematics that may compromise patient satisfaction.

Total knee arthroplasty using functional alignment [FA] aims to restore the patient's prearthritic knee anatomy and native joint kinematics. Early clinical and functional outcome studies have reported promising outcomes in TKA with FA but results of longer term studies have not yet been published.

There are very few prospective studies exploring clinical and radiological outcomes in MA versus FA for TKA. It is possible to improve on previous studies by recording a more comprehensive range of clinical and functional outcome measures, blinding patients and observers recording outcomes of interest, and using longer follow-up times.

Robotic-arm assistance can be used to improve the accuracy of implant positioning. Clinical and functional outcomes should also be correlated to longer-term outcomes to better establish the "safe zone" for functional alignment. The findings of this study will enable an improved understanding of the clinical and functional benefits of FA compared to MA. These outcomes will improve our understanding of the optimal TKA alignment with possible improved outcomes; improved cost-effectiveness by reduced revisions and better patient satisfaction and function; and improved long-term implant survival.

100 patients will be enrolled in a 1:1 ratio between the two treatment groups. Trial patient will be allocated to either the MA TKA ['Control group'] or to the FA TKA ['Investigation group']. Outcomes will be recorded at specific milestones.

ELIGIBILITY:
Inclusion Criteria:

* Patient has symptomatic knee osteoarthritis requiring primary TKA
* Patient and surgeon are in agreement that TKA is the most appropriate treatment
* Patient is fit for surgical intervention following review by surgeon and anaesthetist
* Patient is between 18-80 years of age at time of surgery
* Gender: male and female
* Patient must be capable of giving informed consent and agree to comply with the postoperative review program
* Patient must be a permanent resident in an area accessible to the study site
* Patient must have sufficient postoperative mobility to attend follow-up clinics and allow for radiographs to be taken

Exclusion Criteria:

* Patient is not suitable for routine primary TKA e.g. patient has ligament deficiency that requires a constrained prosthesis
* Patient has bone loss that requires augmentation
* Patient is not medically fit for surgical intervention
* Patient requires revision surgery following previously failed correctional osteotomy or ipsilateral TKA
* Patient is immobile or has another neurological condition affecting musculoskeletal function
* Patient is less than 18 years of age or greater than 80 years of age
* Patient is already enrolled on another concurrent clinical trial
* Patient is unable or unwilling to sign the informed consent form specific to this study
* Patient is unable to attend the follow-up programme
* Patient is non-resident in local area or expected to leave the catchment area postoperatively

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-12-28 (Actual); Primary Completion 2025-02-06 (Actual); Study Completion 2025-02-06 (Actual)

PRIMARY OUTCOMES:
Western Ontario and Mcmaster Universities Arthritis Index (WOMAC) | 2 years post-intervention
  Patient recorded outcome questionnaire evaluating pain, stiffness and disability in affected joint

SECONDARY OUTCOMES:
Lower limb alignment | pre op and 6 weeks post op
  Assessed using Computerised Tomography (CT) scanogram. Measurements of the hip-knee-angle (HKA), medial proximal tibial angle (MPTA), lateral distal femoral angle (LDFA), femoral flexion angle, and posterior tibial slope will be recorded preoperatively and postoperatively
Operating time | interoperative
  Operating time [minutes]
Time to discharge | Documented when participant leaves hospital, an average of 72 -96 hours
  Time to discharge from admission until documented discharge from hospital (hours)
Forgotten Joint Score (FJS) | Pre-op; 6 weeks post-op; 6 months post-op; 1 year post-op; 2 years post-op
  Patient recorded outcome measure via questionnaire. Score cumulative with -100 being best score and 0 being worst score
Oxford Knee Score (OKS) | Pre-op; 6 weeks post-op; 6 months post-op; 1 year post-op; 2 years post-op
  Patient recorded outcome measure via questionnaire. 48 is best score and 0 worst score
Short form health survey of 12 items (SF-12), | Pre-op; 6 weeks post-op; 6 months post-op; 1 year post-op; 2 years post-op
  Patient recorded outcome measure. Questions concerning attitudes to physical and mental heath with 12 questions combined to give overall norm-based values; higher score better, lower score worse.
Knee injury and osteoarthritis outcome score (KOOS) | Pre-op; 6 weeks post-op; 6 months post-op; 1 year post-op; 2 years post-op
  Patient recorded outcome measure via questionnaire. 6 separate domains including pain, stiffness, quality of life, symptoms, and function; each domain creates percentage with overall cumulative percentage achieved; best score 100%
University of California at Los Angeles knee (UCLA) | Pre-op; 6 weeks post-op; 6 months post-op; 1 year post-op; 2 years post-op
  Patient recorded outcome measure via questionnaire. Patient records current level of activity; 10 best possible score, 0 worst possible score
European Quality of Life questionnaire with 5 dimensions for adults (EQ-5D) | Pre-op; 6 weeks post-op; 6 months post-op; 1 year post-op; 2 years post-op
  Patient recorded outcome measure with 5 domains; score -1 to 1, with 1 being best score
Use of mobility aids | during inpatient admission and postoperatively at 6- weeks, 6 months, 1 year and 2 years
  description of any mobility aids used to assist with ambulation; can describe wheelchair, walker, crutches, sticks or no need for any mobility aid
Mobilisation distance | during inpatient admission and postoperatively at 6- weeks, 6 months, 1 year and 2 years
  Mobilisation distance (metres)
Range of movement | inpatient admission and postoperatively at 6 weeks, 6 months, 1 year and 2 years
  Range of movement (degrees) in knee joint
radiosteriometric analysis (RSA) | postoperatively at 2 weeks, 6 weeks, 6 months, 1 year, and 2 years
  Femoral and tibial implant early migration as assessed using RSA
Gait analysis | performed postoperatively at 6 months and 1 year postoperatively
  Walking on an instrumented treadmill with force plates
Complications | during inpatient admission and postoperatively at 6- weeks, 6 months, 1 year and 2 years
  Complications relating to surgery

CONTACTS AND LOCATIONS:
Overall Officials: Fares S Haddad, Study Chair — UCLH
Locations (1):
- University College London Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plan

REFERENCES:
- [Derived] Kayani B, Konan S, Tahmassebi J, Oussedik S, Moriarty PD, Haddad FS. A prospective double-blinded randomised control trial comparing robotic arm-assisted functionally aligned total knee arthroplasty versus robotic arm-assisted mechanically aligned total knee arthroplasty. Trials. 2020 Feb 18;21(1):194. doi: 10.1186/s13063-020-4123-8. PMID 32070406